CLINICAL TRIAL: NCT00041548
Title: Inhaled Nitric Oxide in Neonates With Elevated A-a DO2 Gradients Not Requiring Mechanical Ventilation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CARLW1
Record Dates: First submitted 2002-07-10; First posted 2002-07-11 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Lung Disease; Hypoxemia; Respiratory Acidosis
MeSH Terms: conditions — Lung Diseases; Hypoxia; Acidosis, Respiratory | interventions — Nitric Oxide; Inhalation; Endothelium-Dependent Relaxing Factors; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nitric Oxide for Inhalation
  Interventions: Drug: nitric oxide for inhalation
- 2 (Placebo Comparator): oxygen
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: nitric oxide for inhalation — given at 20 ppm for 1 hour then weaned off over 4 hours
  Other Names: INOmax
  Arms: 1
Drug: Oxygen — given at 20 ppm for one hour, then weaned off over four hours
  Arms: 2

SUMMARY:
The purpose of this pilot study is to evaluate whether administration of nitric oxide (NO)gas by oxygen hood at 20 ppm significantly increases PaO2, as compared to placebo gas (oxygen), within one hour of initiation and with no significant adverse effects.

DETAILED DESCRIPTION:
It is possible that administration of inhaled NO to neonates with abnormal gas exchange earlier, rather than later as a rescue therapy in a moribund state, might accelerate the transition of the circulation from the fetal to neonatal physiology and improve oxygenation. This may in turn decrease the need for mechanical ventilation, its associated morbidity and perhaps even ECMO.

This study is designed as a pilot study to evaluate the physiologic efficacy (rather than effect on clinical outcomes) of NO administered by hood in improving oxygenation of neonates with elevated A-a DO2.

ELIGIBILITY:
Inclusion criteria:

* Gestational age >34 completed weeks (>=35)
* Age <48 hours
* A-a DO2 400 to 600, on two post-ductal arterial blood gases one hour apart, while on 100% O2 by oxygen hood
* Post-ductal arterial access
* Admitted to The University of Alabama Birmingham Regional NICU

Exclusion criteria:

* Cardiac disease (structural disease with right to left or mixing lesions), not including patent ductus arteriosus (PDA) or patent foramen ovale (PFO)
* Rapid deterioration requiring mechanical ventilation before entry into the study
* Major malformations
* Major neurologic or metabolic disorder or other illness leading to hypoventilation and hypercarbia

Max Age: 120 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2002-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
PaO2 level | at baseline, then every hour for 6 hours

SECONDARY OUTCOMES:
Methemoglobin level | at baseline then every hour of treatment
Alveolar-arterial oxygen gradient and ratio | after 1 hour of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Ambalavanan N, El-Ferzli GT, Roane C, Johnson R, Carlo WA. Nitric oxide administration using an oxygen hood: a pilot trial. PLoS One. 2009;4(2):e4312. doi: 10.1371/journal.pone.0004312. Epub 2009 Feb 2. PMID 19183804